CLINICAL TRIAL: NCT03127228
Title: Laser-Assisted Regenerative Surgical Therapy for Peri-implantitis: A Randomized Controlled Clinical Trial
Brief Title: Laser-Assisted Regenerative Surgical Therapy for Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Morita J USA (Unknown)
Responsible Party: Principal Investigator, Chin-Wei Wang, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00124386
Record Dates: First submitted 2017-04-19; First posted 2017-04-25 (Actual); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Peri-Implantitis
Keywords: Laser
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard mechanical debridement (Other): Debridement and surface detoxification of the implant surface and removal of the inflamed tissue with dental scalers.
  Interventions: Other: Standard mechanical debridement
- Er:YAG laser-assisted debridement (Experimental): Debridement and surface detoxification of the implant surface and removal of the inflamed tissue with the aid of the laser treatment.
  Interventions: Other: Standard mechanical debridement; Device: Er:YAG laser-assisted debridement

INTERVENTIONS:
Other: Standard mechanical debridement — Implantoplasty will be performed for peri-implant suprabony defect and infrabony defect will be debrided with dental scalers prior to bone grafting regenerative therapy
Device: Er:YAG laser-assisted debridement — Implantoplasty will be performed for peri-implant suprabony defect and infrabony defect will be debrided with the aid of the laser prior to bone grafting regenerative therapy
  Arms: Er:YAG laser-assisted debridement

SUMMARY:
The purpose of the study is to evaluate if using Erbium-doped yttrium aluminium garnet laser, Erbium YAG laser (Er:YAG) laser could have adjunctive benefits to the conventional standard mechanical debridement to ablate the infected tissue around the dental implant and detoxify the contaminated implant surface for resolving peri-implant infection and enhance bone regeneration of peri-implant defects.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate if using Er:YAG laser could have adjunctive benefits to the conventional standard mechanical debridement to ablate the infected tissue around the dental implant and detoxify the contaminated implant surface for resolving peri-implant infection and enhance bone regeneration of peri-implant defects.

This study involves one center and a double-blinded randomized controlled clinical trial is planned. Twenty-four adult patients in the need of surgical treatment due to peri-implantitis will be included. Six visits are needed for each patient including a 24 week follow-up visit.

Specific Aim 1: To compare the clinical benefit of Er:YAG laser-assisted peri-implant defect debridement and surface detoxification with conventional mechanical debridement for regenerative therapy

Specific Aim 2: To evaluate whether Er:YAG laser-assisted regenerative surgical therapy can decrease bacterial load and alter microbial profile

Specific Aim 3: To analyze whether Er:YAG laser-assisted regenerative surgical therapy can impact the molecular profile of the peri-implant crevicular fluid (PICF) and the stability of the treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects, aged 18 - 85 years
* Physical status according to the American Society of Anesthesiologists (ASA) I or II, which includes patients who are systemically healthy or suffer under mild to moderate, but well controlled systemic diseases.
* Subjects having a minimum of 1 dental implant with peri-implantitis.
* Dental implants with peri-implantitis ≥ 2 threads exposed (infrabony defect) identified on the radiograph and pocket probing depth (PPD) ≥ 5mm, with bleeding on probing (BOP) and/or suppuration (pus)
* The implants are in function for at least 6 months
* Only rough surface implant will be included in this study

Exclusion Criteria:

* Long-term use of antibiotics > 2 weeks in the past two months
* Obvious malpositioning of the dental implants
* Subjects taking medications known to modify bone metabolism (such as bisphosphonates, corticosteroids, Hormone replacement therapy for menopausal women, parathyroid hormone, Denosumab, strontium ranelate)
* Pregnant females or those planning to become pregnant
* Subjects with a history of major diseases, oral cancer, sepsis or those having adverse outcomes to oral procedures in the past, will be excluded
* Mobility of dental implants
* History of alcoholism or drug abuse
* Current smokers
* Diseases of the immune system or any medical condition that may influence the outcome (uncontrolled diabetes (HbA1c >8)
* Uncontrolled systemic disease or condition known to alter bone metabolism, like Osteoporosis, Osteopenia, Hyperparathyroidism, Paget's disease

Premature Exclusion Criteria:

* The researcher believes that it is not the best interest of the subject to stay in the study
* If the subject becomes ineligible to participate based on the exclusion criteria
* If the subject's medical condition requires interventions which preclude involvement in the study (radiation therapy, chemotherapy, etc)
* If the subject does not follow study related instructions
* The study is suspended or canceled.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff (Chin-Wei) Wang, DDS, DMSc, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan School of Dentistry
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aljateeli M, Fu JH, Wang HL. Managing peri-implant bone loss: current understanding. Clin Implant Dent Relat Res. 2012 May;14 Suppl 1:e109-18. doi: 10.1111/j.1708-8208.2011.00387.x. Epub 2011 Oct 10. PMID 21985674
- [Background] Aoki A, Mizutani K, Schwarz F, Sculean A, Yukna RA, Takasaki AA, Romanos GE, Taniguchi Y, Sasaki KM, Zeredo JL, Koshy G, Coluzzi DJ, White JM, Abiko Y, Ishikawa I, Izumi Y. Periodontal and peri-implant wound healing following laser therapy. Periodontol 2000. 2015 Jun;68(1):217-69. doi: 10.1111/prd.12080. PMID 25867988
- [Background] Atieh MA, Alsabeeha NH, Faggion CM Jr, Duncan WJ. The frequency of peri-implant diseases: a systematic review and meta-analysis. J Periodontol. 2013 Nov;84(11):1586-98. doi: 10.1902/jop.2012.120592. Epub 2012 Dec 13. PMID 23237585
- [Background] Claffey N, Clarke E, Polyzois I, Renvert S. Surgical treatment of peri-implantitis. J Clin Periodontol. 2008 Sep;35(8 Suppl):316-32. doi: 10.1111/j.1600-051X.2008.01277.x. PMID 18724859
- [Background] De Bruyn H, Vandeweghe S, Ruyffelaert C, Cosyn J, Sennerby L. Radiographic evaluation of modern oral implants with emphasis on crestal bone level and relevance to peri-implant health. Periodontol 2000. 2013 Jun;62(1):256-70. doi: 10.1111/prd.12004. PMID 23574471
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Fransson C, Lekholm U, Jemt T, Berglundh T. Prevalence of subjects with progressive bone loss at implants. Clin Oral Implants Res. 2005 Aug;16(4):440-6. doi: 10.1111/j.1600-0501.2005.01137.x. PMID 16117768
- [Background] Goncalves F, Zanetti AL, Zanetti RV, Martelli FS, Avila-Campos MJ, Tomazinho LF, Granjeiro JM. Effectiveness of 980-mm diode and 1064-nm extra-long-pulse neodymium-doped yttrium aluminum garnet lasers in implant disinfection. Photomed Laser Surg. 2010 Apr;28(2):273-80. doi: 10.1089/pho.2009.2496. PMID 19811080
- [Background] Jensen MP, Karoly P, O'Riordan EF, Bland F Jr, Burns RS. The subjective experience of acute pain. An assessment of the utility of 10 indices. Clin J Pain. 1989 Jun;5(2):153-9. doi: 10.1097/00002508-198906000-00005. PMID 2520397
- [Background] Kinney JS, Morelli T, Oh M, Braun TM, Ramseier CA, Sugai JV, Giannobile WV. Crevicular fluid biomarkers and periodontal disease progression. J Clin Periodontol. 2014 Feb;41(2):113-120. doi: 10.1111/jcpe.12194. Epub 2013 Dec 12. PMID 24303954
- [Background] Kreisler M, Kohnen W, Marinello C, Gotz H, Duschner H, Jansen B, d'Hoedt B. Bactericidal effect of the Er:YAG laser on dental implant surfaces: an in vitro study. J Periodontol. 2002 Nov;73(11):1292-8. doi: 10.1902/jop.2002.73.11.1292. PMID 12479633
- [Background] Marrone A, Lasserre J, Bercy P, Brecx MC. Prevalence and risk factors for peri-implant disease in Belgian adults. Clin Oral Implants Res. 2013 Aug;24(8):934-40. doi: 10.1111/j.1600-0501.2012.02476.x. Epub 2012 May 3. PMID 22551347
- [Background] Matys J, Dominiak M. Assessment of Pain When Uncovering Implants with Er:YAG Laser or Scalpel for Second Stage Surgery. Adv Clin Exp Med. 2016 Nov-Dec;25(6):1179-1184. doi: 10.17219/acem/62456. PMID 28028971
- [Background] Nevins M, Nevins ML, Yamamoto A, Yoshino T, Ono Y, Wang CW, Kim DM. Use of Er:YAG laser to decontaminate infected dental implant surface in preparation for reestablishment of bone-to-implant contact. Int J Periodontics Restorative Dent. 2014 Jul-Aug;34(4):461-6. doi: 10.11607/prd.2192. PMID 25006763
- [Background] Peri-implant mucositis and peri-implantitis: a current understanding of their diagnoses and clinical implications. J Periodontol. 2013 Apr;84(4):436-43. doi: 10.1902/jop.2013.134001. No abstract available. PMID 23537178
- [Background] Quaranta A, Maida C, Scrascia A, Campus G, Quaranta M. Er:Yag Laser application on titanium implant surfaces contaminated by Porphyromonas gingivalis: an histomorphometric evaluation. Minerva Stomatol. 2009 Jul-Aug;58(7-8):317-30. English, Italian. PMID 19633633
- [Background] Renvert S, Roos-Jansaker AM, Claffey N. Non-surgical treatment of peri-implant mucositis and peri-implantitis: a literature review. J Clin Periodontol. 2008 Sep;35(8 Suppl):305-15. doi: 10.1111/j.1600-051X.2008.01276.x. PMID 18724858
- [Background] Schwarz F, Hegewald A, John G, Sahm N, Becker J. Four-year follow-up of combined surgical therapy of advanced peri-implantitis evaluating two methods of surface decontamination. J Clin Periodontol. 2013 Oct;40(10):962-7. doi: 10.1111/jcpe.12143. Epub 2013 Aug 12. PMID 23931259
- [Background] Schwarz F, Sahm N, Iglhaut G, Becker J. Impact of the method of surface debridement and decontamination on the clinical outcome following combined surgical therapy of peri-implantitis: a randomized controlled clinical study. J Clin Periodontol. 2011 Mar;38(3):276-84. doi: 10.1111/j.1600-051X.2010.01690.x. Epub 2011 Jan 11. PMID 21219392
- [Background] Suarez-Lopez Del Amo F, Yu SH, Wang HL. Non-Surgical Therapy for Peri-Implant Diseases: a Systematic Review. J Oral Maxillofac Res. 2016 Sep 9;7(3):e13. doi: 10.5037/jomr.2016.7313. eCollection 2016 Jul-Sep. PMID 27833738
- [Background] Takasaki AA, Aoki A, Mizutani K, Kikuchi S, Oda S, Ishikawa I. Er:YAG laser therapy for peri-implant infection: a histological study. Lasers Med Sci. 2007 Sep;22(3):143-57. doi: 10.1007/s10103-006-0430-x. Epub 2007 Jan 12. PMID 17219255
- [Background] Wang HL, Garaicoa-Pazmino C, Collins A, Ong HS, Chudri R, Giannobile WV. Protein biomarkers and microbial profiles in peri-implantitis. Clin Oral Implants Res. 2016 Sep;27(9):1129-36. doi: 10.1111/clr.12708. Epub 2015 Oct 1. PMID 26424287
- [Background] Yamamoto A, Tanabe T. Treatment of peri-implantitis around TiUnite-surface implants using Er:YAG laser microexplosions. Int J Periodontics Restorative Dent. 2013 Jan-Feb;33(1):21-30. doi: 10.11607/prd.1593. PMID 23342343
- [Derived] Wang CW, Di Gianfilippo R, Kaciroti N, Ou A, Feng SW, Wang HL. Stability of peri-implantitis surgical reconstructive therapy-a (> 2 years) follow-up of a randomized clinical trial. Clin Oral Investig. 2023 Dec 26;28(1):30. doi: 10.1007/s00784-023-05457-6. PMID 38147180
- [Derived] Wang CW, Ashnagar S, Gianfilippo RD, Arnett M, Kinney J, Wang HL. Laser-assisted regenerative surgical therapy for peri-implantitis: A randomized controlled clinical trial. J Periodontol. 2021 Mar;92(3):378-388. doi: 10.1002/JPER.20-0040. Epub 2020 Aug 25. PMID 32761810

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.41 (13.48) | 66.41 (8.76) | 64.91 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Periodontal Probing Depths (PD)
Description: PD will be measured in millimeters. Change in PD measurements were calculated between baseline and 24 weeks.
Time Frame: Baseline and 24 Week
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement
Number analyzed (Participants) | 12 | 12
Number analyzed (Implants) | 12 | 12
millimeters | 1.85 (1.71) | 2.65 (2.14)

2. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: CAL will be measured in millimeters. Change in subject CAL measurements were calculated between baseline and 24 weeks.
Time Frame: Baseline and 24 Week
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement
Number analyzed (Participants) | 12 | 12
Number analyzed (Implants) | 12 | 12
millimeters | 1.47 (1.76) | 1.90 (2.28)

3. Primary Outcome: Change in Bleeding on Probing (BOP)
Description: BOP will be measured dichotomously as 0 or 1. Score 0=no bleeding present Score 1=bleeding present Change in subject BOP score was calculated between baseline and 24 weeks and reported as percent of sites with BOP.
Time Frame: Baseline and 24 Week
Measure: Mean (Standard Deviation); unit: percentage of sites with BOP
Units Other Than Participants: Implants
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement
Number analyzed (Participants) | 12 | 12
Number analyzed (Implants) | 12 | 12
percentage of sites with BOP | -0.39 (0.55) | -0.31 (0.62)

4. Primary Outcome: Change in Radiographic Bone Fill (RBF)
Description: Peri-implant bony defect change will be measured compared to baseline. Participants' standardized radiographs were used to determine bone level changes between baseline and 24 weeks.
Time Frame: Baseline and 24 Week
Measure: Mean (Standard Deviation); unit: Millimeters
Units Other Than Participants: Implants
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement
Number analyzed (Participants) | 12 | 12
Number analyzed (Implants) | 12 | 12
Millimeters | 1.08 (1.04) | 1.27 (1.14)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The methods for gathering adverse events included a medical and dental history review at each study visit and an oral exam at each study visit. In addition, participants self-reported any adverse events.
Arm/Group | Standard Mechanical Debridement | Er:YAG Laser-assisted Debridement
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Mechanical Debridement (N=12) | Er:YAG Laser-assisted Debridement (N=12)
Sinus Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — During medical/dental history update participant reported having a sinus tract infection. Dispensed antibiotics and referred participant to their primary care physician.
Tooth pain (General disorders) | 1 (1) | 0 (0) — Participant reported tooth pain in lower right quadrant of his mouth. This was a non-study tooth. Participant was referred to his general dentist for care.
Flu (Infections and infestations) | 1 (1) | 0 (0) — Participant reported having the flu and currently taking antibiotics.
Jaw discomfort (General disorders) | 1 (1) | 0 (0) — Participant reported having jaw discomfort in both of his jaw joints. Participant was currently being treated by his general dentist.
Broken filling (General disorders) | 0 (0) | 1 (1) — Participant reported having a broken filling on a non-study tooth. Participant had an appointment scheduled with their general dentist for care.
Shoulder Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — During medical and dental history update the participant reported to have fallen on her shoulder and went to see her primary care physician for treatment.
Fistula (Infections and infestations) | 1 (1) | 0 (0) — Participant reported having a "water bubble" on the inside of his lower left molar. Upon examination it was determined that the participant could have a root canal infection. Participant was referred to a root canal specialist for treatment.
Ulcer on ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) — During the oral exam it was noticed that the participant had an ulcer on his right ear. Participant was referred to this primary care physician for care.
Residual suture (General disorders) | 0 (0) | 1 (1) — Participant reported that there was a residual suture in his mouth. Suture was removed.
Shingles (Immune system disorders) | 0 (0) | 1 (1) — Participant reported that he had shingles and was being treated by his primary care physician.
Crown off (General disorders) | 0 (0) | 1 (1) — Participant reported that the crown fell off of his tooth (non-study tooth). Participant was referred to general dentist for treatment.
Type 2 Diabetes (Immune system disorders) | 1 (1) | 0 (0) — During medical/dental history review the participant reported to have recently been diagnosed with type 2 diabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03127228/Prot_SAP_000.pdf